CLINICAL TRIAL: NCT07099222
Title: Extended Duration of Peripheral Nerve Blocks With Low, Non-weight-based Adjuncts of Dexamethasone and Dexmedetomidine Compared to Dexamethasone Alone in Orthopedic Surgery: A Prospective, Single-blind, Randomized Controlled Trial
Brief Title: Efficacy of Non-weight Based, Low Dose Dex-Dex Adjuncts in Prolonging Peripheral Nerve Blocks
Acronym: Dex-Dex PNB
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ronald Tang, MD, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00004763
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Nausea and Vomiting, Postoperative; Dizziness; Constipation; Duration of Response; Narcotics Consumption; Pain After Surgery
Keywords: Peripheral nerve block; PNB; Dex-Dex; Adjuncts; Dexmedetomidine; Dexamethasone; Extended Nerve Block; Additive; Prolonged Nerve Block; Dex; Steroid; Precedex; Decadron; Brachial Plexus; Sciatic; Femoral; Popliteal; Saphenous; Adductor Canal
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Dizziness; Constipation | interventions — Dexmedetomidine; Dexamethasone; Ropivacaine

STUDY DESIGN:
Intervention Model Description: There will be a control group and a study group. A pre-determined order will be made for assignment into groups. There will be a separate predetermined randomization for patients undergoing shoulder surgery and patients undergoing foot/ankle surgery to help evenly distribute the number of participants assigned to the control and study groups in each subset. The control groups for both shoulder and foot/ankle surgery will receive Ropivacaine with Dexamethasone injection for their peripheral nerve block(s) in the same concentration. The study groups will receive nerve blocks containing Ropivacaine with Dexamethasone and Dexmedetomidine in the same concentration.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group: nerve blocks containing Ropivacaine and Dexamethasone only (Experimental): Ropivicaine peripheral nerve block solution with 4mg Dexamethasone adjunct
  Interventions: Drug: Ropivacaine with low, non weight based Dexamethasone additive
- Study Group: nerve blocks containing Ropivacaine, Dexamethasone, and Dexmedetomidine (Experimental): Ropivacaine local anesthetic solution with 4mg Dexamethasone AND 25mcg Dexmedetomidine added
  Interventions: Drug: Low, non-weight based dose of Dexamethasone and Dexmedetomidine in peripheral nerve blocks

INTERVENTIONS:
Drug: Low, non-weight based dose of Dexamethasone and Dexmedetomidine in peripheral nerve blocks — Low, non-weight based dose of Dexamethasone and Dexmedetomidine adjunct with Ropivacaine (local anesthetic) for use in peripheral nerve blocks to look for synergistic effects of the combination in extending the duration of the block while limiting any potential side effects of each additive.
  Other Names: Dexamethasone and Dexmedetomidine
  Arms: Study Group: nerve blocks containing Ropivacaine, Dexamethasone, and Dexmedetomidine
Drug: Ropivacaine with low, non weight based Dexamethasone additive — Very accepted, standard peripheral nerve block with steroid adjunct solution used to increase the duration of local anesthetic by 4-6hrs.
  Other Names: Ropivacaine and Dexamethasone
  Arms: Control Group: nerve blocks containing Ropivacaine and Dexamethasone only

SUMMARY:
The goal of this clinical study is to improve upon the standard practice of utilizing nerve blocks to enhance the satisfaction of patients undergoing shoulder, or foot and ankle surgery regarding their quality of pain control, the duration of their nerve blocks, as well as the avoidance of opioid medications and subsequently their undesirable side effects. The researchers hypothesize that dexmedetomidine and dexamethasone (Dex-Dex) will work synergistically as adjuncts in a low, non-weight based formula. This would allow the investigators to improve patient satisfaction by providing them with a superior means of pain control that is longer in duration with a decreased probability of unwanted side effects.

The proposed clinical study will be a prospective, randomized control trial.

DETAILED DESCRIPTION:
The standard practice for anesthesia in non-weight-bearing orthopedic foot and ankle surgery is to offer the patient popliteal (sciatic nerve) and saphenous (distal branch of femoral nerve) peripheral nerve blocks for postoperative pain control to minimize opioid requirements. Similarly, supraclavicular nerve blocks that decrease painful stimuli transmission through the brachial plexus are offered to patients undergoing shoulder joint procedures. For these peripheral nerve blocks, it is routine to use dexamethasone (glucocorticoid) as an additive in the local anesthetic injection which can prolong the local anesthetic effect of the blocks by 4-8 hours with minimal side effects observed and no dose-response relationship with perineural injection doses of 4, 8, 10, and 12mg. Though the precise mechanism of action has not been fully understood, it is largely believed that perineural injection of dexamethasone increases the effects of local anesthetics at least in part due to vasoconstriction.

Current literature suggests that 1-2 mcg/kg of dexmedetomidine will also prolong the peripheral nerve blocks but consistent utilization thus far has been limited by side-effects of higher, more efficacious doses. The potential dose-dependent side effects associated with the use of perineural dexmedetomidine include bradycardia, hypotension, and excessive sedation. There are minimal to no side-effects observed when perineural dexmedetomidine doses are kept below 1 mcg/kg. However, its effects on prolonging nerve blocks are not significant until the dose is increased to 1.5 mcg/kg where the nerve block is extended roughly 4-8 hours, similar to using dexamethasone as an adjunct. At doses greater than 2 mcg/kg, however, the nerve block can last up to 2-3 days but at the tradeoff of increased perioperative bradycardia and hypotension from presumed systemic absorption and dexmedetomidine's highly selective α2 agonist effects. Another study showed that when a low, non-weight-based dose of 50 mcg of dexmedetomidine was used in adults weighing over 50 kg, the duration of analgesia was improved, but its effects were less than 8 mg of dexamethasone as an adjunct, and the improvement of the duration of blockade at this low dose of dexmedetomidine was not significant. When both dexamethasone and dexmedetomidine were utilized as intravenous adjuncts administered at the time of performing the nerve blocks instead of in the perineural injection, Maagaard et al. discovered that dexamethasone improved the duration of analgesia of popliteal and saphenous nerve blocks in patients undergoing foot and ankle surgeries with or without dexmedetomidine. These findings support the theory that dexmedetomidine's local effects at the site of the injection, as opposed to its systemic analgesic effects on α2 receptors in the central nervous system, may be predominantly responsible for its role as an adjunct in prolonging the effects of local anesthetics in peripheral nerve blocks. The theory is also supported by Brummett et al and their findings that the analgesic effects of dexmedetomidine as an adjunct could not be reversed by an α2 receptor antagonist given systemically.

This study aims to determine a safe and effective approach for using dexamethasone and dexmedetomidine in combination using low, non-weight based (NWB) doses of both adjuncts. The researchers plan to track the duration of the blocks for 7 days postoperatively as well as any unwanted side effects in the post-anesthesia care unit including: hypotension, bradycardia, oversedation, and respiratory depression. The research team will contact subjects by email and rely on daily participant surveys (REDCap Survey POD #0) submitted electronically to provide subjective feedback on block duration and postoperative pain for 7 days using the PROMIS pain scale within the survey. Participants will also report pain medication usage for the same time frame including both opioid and non-opioid medications. Side effects in the post anesthesia care unit (PACU) will be documented by PACU nurses using the POSS sedation scale and comparing vital signs such as heart rate and blood pressure at 15- and 30-minute intervals to pre-operation recordings. Subjects might receive a phone call reminder to complete the daily surveys after their surgery, or if the research team notices that they have not completed the surveys on time.

Preliminary data has been very promising. The investigator's facility has thus far declined the use of liposomal bupivacaine, which has limited the ability to offer the patients peripheral nerve blocks lasting greater than 24 hours. Therefore, to extend the length of our peripheral nerve blocks the research team added both 4 mg dexamethasone and 50 mcg dexmedetomidine to 30 ml of 0.5% ropivacaine for lower extremity blocks for patients that would benefit from a prolonged nerve block for postoperative pain. The roughly 31.5 ml solution is then split evenly between the popliteal and saphenous nerve blocks. The investigators observed that these blocks frequently extended the duration of the block to 2-5 days compared to the standard 20-24 hours normally observed with dexamethasone adjunct alone. Similarly, the exact same additives (4 mg dexamethasone and 50 mcg dexmedetomidine) have been added to 15 ml of 0.5% Ropivacaine for shoulder procedures with similar observations noted of increased duration. This posed a research question that the investigators wishe to investigate further that compares their usual practice of blocks with ropivacaine and dexamethasone alone to blocks utilizing both dexamethasone and dexmedetomidine as adjuncts. The investigators chose the dexmedetomidine dose in combination with their inclusion criteria of adults weighing more than 50 kg so that the patients in this study will not receive a dexmedetomidine adjunct dose that is greater than 1 mcg/kg.

For the initial research the investigators plan on recruiting patients who are undergoing foot and ankle surgery who are not expected to participate in weight-bearing physical rehabilitation immediately after surgery and that would benefit from a potential multi-day nerve block for primary pain management. The investigators also plan on recruiting patients undergoing extensive shoulder surgery such as total shoulder arthroplasty and rotator cuff repairs because these procedures tend to have higher observed post-operative pain associated and the patients are not expected to participate in active rehabilitation immediately after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (18 years and older but less than 75)
* Speaks and understands English.
* Capable of performing all activities of daily living independently
* Normal development for age and without cognitive impairment
* Weight over 50 kg
* Undergoing scheduled, elective foot, ankle, and shoulder surgery
* Patient is not expected to perform weight-bearing rehabilitation post-op for 1 week.
* Regular access to the internet

Exclusion Criteria:

* Under 18 or older than 75 years of age
* Pregnancy
* Known allergy to local anesthetics including lidocaine and ropivacaine.
* Known allergy to glucocorticoid steroids or necessary abstinence for medical reasons.
* Known allergy to dexmedetomidine or other α2 agonist derivatives.
* Severe organ dysfunction: end-stage renal disease, liver failure
* Severe psychiatric disease that alters sense of reality and interferes with pain perception.
* Severe cognitive impairment that interferes with pain perception
* Chronic opioid use, alcohol abuse, or any other substance abuse
* Urgent/emergent procedure
* Emergency return to OR after initial surgery
* Infection at block or surgical site
* Hemodynamic instability preoperatively
* Hemodynamic instability during surgery affects timely extubating at the end of surgery.
* Failed nerve blocks that did not end up blocking the nerves as intended, or inadequate nerve blocks requiring repeat rescue blocks in PACU.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral Nerve Block Duration | 0-7 days
  Using automated daily emailed patient surveys to assess for the duration of the peripheral nerve block.
Post-operative pain scores | 0-7 days
  Postoperative pain scores based on the Patient-Reported Outcomes Measurement Information System (PROMIS) numeric rating scale for pain intensity with response scores from 0 (no pain) to 10 (pain as bad as it can be) are to be reported daily by the participant for 7 days after surgery. Therefore, a higher score on the scale would indicate a worse outcome in terms of pain experienced by the participant.
Pain medicine (opioid and non-opioid) consumption post-operatively | 0-7 days
  Opioid and non-opioid pain medication consumption postoperatively, reported daily by the participant for 7 days

SECONDARY OUTCOMES:
Post-opertive side effects | 0-7 days
  Measuring any reduction in opioid use side effects in the study group as a result of increased block duration leading to less opioid use for breakthrough pain. These side effects measured include: nausea, vomiting, lightheadedness, dizziness, and constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Tang, MD, Principal Investigator — University of Arizona - Banner Health
Locations (1):
- Banner - University Medical Center South, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical researchers may contact the principal investigator (Ronald Tang, MD) to request the raw data for the study. All shared data will be void of personal identifiers. Sharing of data will be granted on a case by case basis determined by the credentials of the requesting researcher and necessity for requesting the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results.
Access Criteria: Researchers studying the effects of Dexmedetomidine and Dexamethasone may request access to the IPD and supporting information. The principal investigator will ultimately decide if criteria is met for data to be shared. In addition, a data sharing agreement may need to be signed on accordance with the University of Arizona and Banner University Medical Center policies.

REFERENCES:
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400
- [Background] Andersen JH, Karlsen A, Geisler A, Jaeger P, Grevstad U, Dahl JB, Mathiesen O. Alpha2 -receptor agonists as adjuvants for brachial plexus nerve blocks-A systematic review with meta-analyses. Acta Anaesthesiol Scand. 2022 Feb;66(2):186-206. doi: 10.1111/aas.14002. Epub 2021 Dec 21. PMID 34811722
- [Background] Chen Z, Liu Z, Feng C, Jin Y, Zhao X. Dexmedetomidine as an Adjuvant in Peripheral Nerve Block. Drug Des Devel Ther. 2023 May 17;17:1463-1484. doi: 10.2147/DDDT.S405294. eCollection 2023. PMID 37220544
- [Background] Singh N, Gupta S, Kathuria S. Dexmedetomidine vs dexamethasone as an adjuvant to 0.5% ropivacaine in ultrasound-guided supraclavicular brachial plexus block. J Anaesthesiol Clin Pharmacol. 2020 Apr-Jun;36(2):238-243. doi: 10.4103/joacp.JOACP_176_19. Epub 2020 Jun 15. PMID 33013041
- [Background] Venkatraman R, Pushparani A, Karthik K, Nandhini P. Comparison of morphine, dexmedetomidine and dexamethasone as an adjuvant to ropivacaine in ultrasound-guided supraclavicular brachial plexus block for postoperative analgesia-a randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2021 Jan-Mar;37(1):102-107. doi: 10.4103/joacp.JOACP_70_19. Epub 2021 Apr 10. PMID 34103832
- [Background] Maagaard M, Funder KS, Schou NK, Penny JO, Toquer P, Laigaard J, Stormholt ER, Norskov AK, Jaeger P, Andersen JH, Mathiesen O. Combined Dexamethasone and Dexmedetomidine as Adjuncts to Popliteal and Saphenous Nerve Blocks in Patients Undergoing Surgery of the Foot or Ankle: A Randomized, Blinded, Placebo-controlled Clinical Trial. Anesthesiology. 2024 Jun 1;140(6):1165-1175. doi: 10.1097/ALN.0000000000004977. PMID 38489226
- [Background] Brummett CM, Amodeo FS, Janda AM, Padda AK, Lydic R. Perineural dexmedetomidine provides an increased duration of analgesia to a thermal stimulus when compared with a systemic control in a rat sciatic nerve block. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):427-31. doi: 10.1097/AAP.0b013e3181ef4cf0. PMID 20814283
- [Background] Desai N, Albrecht E, El-Boghdadly K. Perineural adjuncts for peripheral nerve block. BJA Educ. 2019 Sep;19(9):276-282. doi: 10.1016/j.bjae.2019.05.001. Epub 2019 Jul 6. No abstract available. PMID 33456903
- [Background] Obayah GM, Refaie A, Aboushanab O, Ibraheem N, Abdelazees M. Addition of dexmedetomidine to bupivacaine for greater palatine nerve block prolongs postoperative analgesia after cleft palate repair. Eur J Anaesthesiol. 2010 Mar;27(3):280-4. doi: 10.1097/EJA.0b013e3283347c15. PMID 19935071
- [Background] Iyengar SS, Pangotra A, Abhishek K, Sinha N, Rao NS, Singh VK, Prakash J. The Comparison of Dexmedetomidine to Dexamethasone as Adjuvants to Bupivacaine in Ultrasound-Guided Infraclavicular Brachial Plexus Block in Upper Limb Surgeries. Cureus. 2023 Jul 10;15(7):e41668. doi: 10.7759/cureus.41668. eCollection 2023 Jul. PMID 37575723
- [Background] Schubert AK, Seneviratne V, Stolz J, Wiesmann T, Wulf H, Eberhart L, Dinges HC. The effect of adjuvants added to local anaesthetics for single-injection upper extremity peripheral regional anaesthesia: A systematic review with network meta-analysis of randomised trials. Eur J Anaesthesiol. 2023 Sep 1;40(9):672-690. doi: 10.1097/EJA.0000000000001860. Epub 2023 Jun 19. PMID 37337656
- [Background] Wei XM, Liu Z, Lv LC, Wu GH, Sun PY, Gu CP, Shi PC. Comparison of dexmedetomidine and dexamethasone as adjuvants to the ultrasound-guided interscalene nerve block in arthroscopic shoulder surgery: a systematic review and Bayesian network meta-analysis of randomized controlled trials. Front Med (Lausanne). 2023 Jun 16;10:1159216. doi: 10.3389/fmed.2023.1159216. eCollection 2023. PMID 37396910
- [Background] Edinoff AN, Houk GM, Patil S, Bangalore Siddaiah H, Kaye AJ, Iyengar PS, Cornett EM, Imani F, Mahmoudi K, Kaye AM, Urman RD, Kaye AD. Adjuvant Drugs for Peripheral Nerve Blocks: The Role of Alpha-2 Agonists, Dexamethasone, Midazolam, and Non-steroidal Anti-inflammatory Drugs. Anesth Pain Med. 2021 Jul 4;11(3):e117197. doi: 10.5812/aapm.117197. eCollection 2021 Jun. PMID 34540647
- [Background] Brummett CM, Hong EK, Janda AM, Amodeo FS, Lydic R. Perineural dexmedetomidine added to ropivacaine for sciatic nerve block in rats prolongs the duration of analgesia by blocking the hyperpolarization-activated cation current. Anesthesiology. 2011 Oct;115(4):836-43. doi: 10.1097/ALN.0b013e318221fcc9. PMID 21666435
- [Background] Marhofer P, Brummett CM. Safety and efficiency of dexmedetomidine as adjuvant to local anesthetics. Curr Opin Anaesthesiol. 2016 Oct;29(5):632-7. doi: 10.1097/ACO.0000000000000364. PMID 27258154
- [Background] Chen BS, Peng H, Wu SN. Dexmedetomidine, an alpha2-adrenergic agonist, inhibits neuronal delayed-rectifier potassium current and sodium current. Br J Anaesth. 2009 Aug;103(2):244-54. doi: 10.1093/bja/aep107. Epub 2009 Jun 20. PMID 19542547
- [Background] Reddy BS, Gaude YK, Vaidya S, Kini GK, Budania LS, Eeshwar MV. Effect of dexmedetomidine on characteristics of ultrasound-guided supraclavicular brachial plexus block with levobupivacaine-A prospective double-blind randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2021 Jul-Sep;37(3):371-377. doi: 10.4103/joacp.JOACP_289_18. Epub 2021 Oct 12. PMID 34759546
- [Background] Jung HS, Seo KH, Kang JH, Jeong JY, Kim YS, Han NR. Optimal dose of perineural dexmedetomidine for interscalene brachial plexus block to control postoperative pain in patients undergoing arthroscopic shoulder surgery: A prospective, double-blind, randomized controlled study. Medicine (Baltimore). 2018 Apr;97(16):e0440. doi: 10.1097/MD.0000000000010440. PMID 29668608